CLINICAL TRIAL: NCT06290726
Title: Long-term Outcomes of Active Vaccination Against de Novo Hepatitis B Among Pediatric Recipients of Living Donor Liver Transplantations With Anti-HBc (+) Grafts
Brief Title: Long-term Outcomes of Living Donor Liver Transplantations With Anti-HBc (+) Grafts in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chih-Che Lin, Professor, Chang Gung Memorial Hospital
Other Study IDs: 202001927B0
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Living Donor Liver Transplantations With Anti-HBc (+) Grafts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- living donor liver transplantations with anti-HBc (+) grafts: No intervention(s) had been administered.
- living donor liver transplantations with anti-HBc (-) grafts: No intervention(s) had been administered.

SUMMARY:
The goal of this observational study is to compare in anti-HBc (+) grafts/ anti-HBc (-) grafts. The main question it aims to answer is the long-term efficacy of active vaccination and graft/patient outcomes of anti-HBc (+) grafts have yet to be comprehensively investigated. Researchers will compare anti-HBc (+) grafts/ anti-HBc (-) to see if it would affect the long-term survival.

DETAILED DESCRIPTION:
A particular strength of the present study is in the inclusion of a consecutive cohort of pediatric LDLT recipients with long-term details of follow-up, although there are several limitations. First, this was a retrospective study conducted at a single medical center. Second, the HBV prophylaxis changed from lamivudine to entecavir in 2008, therefore investigators were unable to evaluate the risk of developing lamivudine resistance. In addition, the DNA level data for the donor and graft tissues were lacking. Lastly, this study was conducted in an area with a high prevalence of anti-HBc positivity.

ELIGIBILITY:
Inclusion Criteria:

- consecutive pediatric LDLT recipients.

Exclusion Criteria:

* Adult LDLT recipients

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The consecutive pediatric LDLT recipients enrolled at a tertiary medical center from February 2002 to February 2016, with follow-up to December 2023.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2002-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
Long-term survival in pediatric recipients of living donor liver transplantations with anti-HBc (+) grafts | Feb. 2002-Feb.2016
  Investigation of the Long-term survival in pediatric recipients of living donor liver transplantations with anti-HBc (+) grafts

IPD SHARING:
Plan to Share IPD: No